CLINICAL TRIAL: NCT02869191
Title: Blood Cultures's Profitability in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Susana Arias Rivera, Registered Nurse, Hospital Universitario Getafe
Other Study IDs: blood cultures
Record Dates: First submitted 2012-07-18; First posted 2016-08-16 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- blood cultures: Admitted patients in critical care who need blood cultures
- blood cultures Getafe: Data collection of patients included in study

SUMMARY:
The purpose of this study is to assess the blood cultures' profitability in intensive care unit and create a validated prediction rule for extractioning in critical patients.

DETAILED DESCRIPTION:
Implementing a predictive rule blood cultures to determine the probability of positive or negative result, improving the profitability of the diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been extracted blood culture sample

Exclusion Criteria:

* Under-aged, pregnants, Major burns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admitted patients in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Percentage of positive, negative and contaminated blood cultures | 2 years

SECONDARY OUTCOMES:
Percentage of positive, negative and contaminated blood cultures after training program | 9 months
  the effect of applying a blood culture extraction protocol is measured

OTHER OUTCOMES:
Contamination rates of blood cultures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susana Arias, RN, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hopsital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No